CLINICAL TRIAL: NCT00663156
Title: A Prospective Study of Autologous Fat Grafting for Breast Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Scott L. Spear, M.D., Chief Plastic Surgery, Georgetown University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4359-617
Record Dates: First submitted 2008-04-01; First posted 2008-04-22 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Breast Augmentation; Fat Grafting
Keywords: lipoaugmentation; breast augmentation; fat grafting; liposuction; lipoinfiltration; Spear; breast implants; ASERF; Lipivage; Baker; harvest; autologous; Georgetown
MeSH Terms: interventions — Breast Implants; Idoxuridine; Lipectomy

ARMS (2):
- subject (Experimental): 10 subjects receiving breast augmentation with fat grafting
  Interventions: Procedure: Liposuction, fat grafting
- control (Other): 10 control will have breast augmentation using breast implants
  Interventions: Procedure: breast implants

INTERVENTIONS:
Procedure: breast implants — patients will have breast augmentation using implants
  Other Names: Allergan; Mentor
  Arms: control
Procedure: Liposuction, fat grafting — Autologous fat will be harvested from the body (typically the abdomen or thighs) using syringe aspiration techniques and then infiltrated into the subcutaneous tissue around the breast as well as between the breast and the underlying musculature using blunt cannulas. These procedures will be done in an outpatient surgery setting in the Georgetown University Hospital under general anesthesia and sterile conditions.
  Other Names: Lipovage; Vectra 3-D
  Arms: subject

SUMMARY:
This research study is to evaluate the natural history of fat transplanted from a person's body to their breasts. We are seeking a natural, safe, and effective alternative to breast implants. Patients will undergo liposuction of their body followed by infiltration of this harvested fat around their breasts. The study protocol will involve preoperative and postoperative photographs, mammograms, and MRI to look for changes in the breast shape and size, as well as any internal changes in the breast tissue.

DETAILED DESCRIPTION:
The current standard for breast augmentation involves placement of an implant. Although implants are safe, they are foreign bodies and thus have inherent risks including infection, failure, malposition, etc. In order to avoid the inherent risks of an implanted device, some surgeons and patients have elected to proceed with breast augmentation from autologous tissue. Early reports of autologous fat transplantation to the breasts were successful, but increases in breast volume were modest (Bircoll, 1987). There were also hypothetical concerns about changes in the breast tissue that would interfere with mammographic screening for breast cancer.

Spear et al (2005) performed autologous fat transplantation to reconstructed breasts in 37 patients with 2-dimensional photographic evidence of improved breast shape and volume suggesting that this technique can be effectively performed. However, these patients had all received mastectomies so mammographic screening was not indicated. Coleman and Saboeiro (2007) performed autologous fat transplantation to the breasts in 17 patients. Fifteen of the 17 patients received post-operative mammograms, 7 (47%) of which were abnormal. However, none of these abnormal findings interfered with cancer screening. Furthermore, 2 patients in the study did develop breast cancer which was successfully detected by mammography. Other studies have confirmed the ability to differentiate benign from malignant findings on mammogram after autologous fat transplantation. Pulagam et al (2006) reported long term (10 and 8 year) findings on 2 patients that underwent autologous fat transplantation to the breasts. Mammography and ultrasound were used to differentiate benign from malignant appearing calcifications. Some authors have speculated that autologous fat transplantation to the breast would lead to mammographic changes similar to routine breast procedures such as breast reduction and mastopexy (Coleman and Saboeiro, 2007).

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years old
* willing to have mammogram, MRI, and photographs
* willing to follow study requirements and sign informed consent
* no previous breast surgeries
* must reside within 50 miles of the Washington, D.C. Metropolitan area

Exclusion Criteria:

* pregnant or nursing
* existing breast cancer
* advanced fibrocystic disease
* protease inhibitors
* any condition leading to surgical risk
* any disease known to affect wound healing
* abscess or infection in the body
* incompatible psychological factors

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness will be evaluated by comparing breast volume pre-operatively and at 1 year post-operatively using 3-dimensional picture imaging to obtain objective volume measurements. | One year post-op

SECONDARY OUTCOMES:
Patients will be evaluated by mammogram, MRI, and 3-D photography to monitor for breast tissue abnormalities and measure increase in volume | one year

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Spear, MD, Principal Investigator — Georgetown University hospital
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States